CLINICAL TRIAL: NCT06553222
Title: Minimally Invasive Non-surgical Therapy With or Without Injectable Bone Putty in Treating Intra-bony Periodontal Defects (Randomized Controlled Clinical Trial)
Brief Title: Minimally Invasive Non-surgical Therapy With or Without Injectable Bone Putty
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Hagar Ahmed Saad, Investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AUAREC20240007-5
Record Dates: First submitted 2024-08-11; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Periodontal Bone Defects
Keywords: periodontal bone defect -bone putty -infrabony defect

STUDY DESIGN:
Intervention Model Description: 2 parallel groups study group - The interventional group where minimally invasive debridement flap and a putty bone graft is tested and the Control group - where minimally invasive debridement flap is performed without graft
Who Masked: Outcomes Assessor
Masking Description: the outcome assessor will assess the bone gain (Radiographic) and Clinical attachment level (clinical) in both groups. the assessor is blinded whether a graft was loaded at the time of surgery
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): Participants receives Injectable bone putty - Minimally invasive debridement periodontal flap plus putty bone graft in three osseous wall defect
  Interventions: Biological: Putty bone - Tricalcium phosphate with Collagen gel
- Control group (Placebo Comparator): - Participants receive No graft (No drug) Minimally invasive debridement periodontal flap
  Interventions: Biological: Putty bone - Tricalcium phosphate with Collagen gel

INTERVENTIONS:
Biological: Putty bone - Tricalcium phosphate with Collagen gel — Minimally invasive debridement periodontal flap and Bone graft placement to augment the lost alveolar bone

SUMMARY:
• All periodontitis patients with infra bony pockets to be included in this study will diagnosed as having stage III periodontitis with probing pocket depth (PPD) ≥ 6 mm, and clinical attachment loss (CAL) ≥ 5mm will be treated by minimally invasive non-surgical therapy or by injectable bone putty

DETAILED DESCRIPTION:
The present study will be designed as a randomized controlled clinical and radiographic. The study will be carried out on stage III grade (B) periodontitis patients with intra-bony defects. Those patients will be selected from the outpatient clinics of the Department of Oral Medicine and Periodontology, Faculty of Dental Medicine, Al-Azhar University, Assiut branch.

The study has bee approved by the ethical committee, Faculty of Dental medicine, Al-Azhar University, Assiut branch.

2. All patients will be fully informed about the study's nature and the possible risks of the study procedures; they sign the consent form before the work.

ELIGIBILITY:
Inclusion Criteria:

* • All periodontitis patients to be included in this study should be diagnosed as having stage III periodontitis with probing pocket depth (PPD) ≥ 6 mm, and clinical attachment loss (CAL) ≥ 5mm.

  * 2- or 3-wall intra-bony interproximal defect with depth ≥3 mm, a width of ≥3 mm at its most coronal part and 45-55-degree angulation will be selected in order to reduce defect variability
  * All patients will be free from any systemic diseases according to the American Dental Academy general guidelines for referring dental patients to specialists and other care settings.

Exclusion Criteria:

• Any patients with any systemic condition that contraindicate any surgical intervention

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-04 (Estimated); Primary Completion 2025-10-04 (Estimated); Study Completion 2025-12-04 (Estimated)

PRIMARY OUTCOMES:
Primary outcome | measured at 6 and 12 months postoperative
  measurement (mm) in alveolar bone gain